CLINICAL TRIAL: NCT06578013
Title: Effect of Acupressure-Ice Message on Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Ashraf Abd El-Ghany, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005306
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure ice massage + pelvic rocking exercises (Experimental): It will include 25 participants suffering from primary dysmenorrhea who will receive acupressure ice massage on SP6 and L14 acupoints, 10 minutes on each point for 20 minutes each session, 5 sessions per cycle (through the 5 days before menstruation) for 3 consecutive menstrual cycles, in addition to pelvic rocking exercises, 15 minute/session, 3 times /week, for 3 successive menstrual cycles.
  Interventions: Other: acupressure ice massage; Other: pelvic rocking exercises
- pelvic rocking exercises (Active Comparator): It will include 25 participants suffering from primary dysmenorrhea, who will perform pelvic rocking exercises only, 15 minutes/session, 3 times /week, for 3 successive menstrual cycles.
  Interventions: Other: pelvic rocking exercises

INTERVENTIONS:
Other: acupressure ice massage — * It will be used for participants in group (A), 2 cm diameter circular ice pieces will be placed inside plastic bags and covered with a thin gauze to prevent moisture transmission and direct ice contact with the skin to apply ice massage.
  * Ice massage will carried out rotationally each 1 minute (30 seconds clockwise and 30 seconds counterclockwise) on L14 point for 10 minutes and on SP6 point for another 10 minutes.
  Arms: acupressure ice massage + pelvic rocking exercises
Other: pelvic rocking exercises — * Pelvic rocking exercise will be used for all participants in both groups (A & B).
  * Each participant will be encouraged to lie down on her back on matrix with a pillow under head then bend her knees and keep her foot flat on the floor and place one hand under curve of her back and the other hand on the top of. her abdomen then tighten buttocks and abdominal muscles simultaneously. After that each participant will be encouraged to inhale and hold (1-2-3-4) then exhale and hold 4-3-2-1 then relax muscles and feel her back flat on the underneath hand. Finally, each participant will be encouraged to repeat the last two steps about 10 times each session.
  * The exercise will be repeated for 15times/ session, 3 times /week, for 3 successive menstrual cycles.

SUMMARY:
This study will be conducted to determine the effect of acupressure ice massage on primary dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is considered the most common gynecological complaint by young women and affects approximately 60-80% of the female population. Around 8-18% of that population report intense discomfort, causing absenteeism in several daily activities while suffering pain.

Analgesics are considered the first line of treatment, but they are known for their undesirable effects such as renal, cardiovascular and gastrointestinal complications that can negatively affect patients' health. Physical therapy has alternative techniques that assist in analgesia in a practical and effective way; among them is acupressure and cryo therapy.

The effect of application of ice on the skin has a direct action on neurons and pain receptors, lowering the speed and the number of nerve impulses. This effect is due to its action on the gate control of pain mechanism, leading to the release of endorphins and enkephalins that are pain-relieving substances.

It was proved from previous studies that using ice massage on L14 or SP6 points reduce pain intensity in females suffering from PD. So, further studies are needed to investigate the effect of acupressure ice massage not only on pain intensity but also on other symptoms severity and quality of life of females suffering from PD. Therefore, this study will be conducted for this issue which will be of valuable benefits for medical service organization and increase body of knowledge of physical therapy in scientific field.

ELIGIBILITY:
Inclusion Criteria:

* Fifty adolescents' females who are clinically diagnosed as primary dysmenorrhea.
* Their ages will be ranged from 17-25 years old.
* Their BMI will be less than 30 kg/m².
* All of them are virgin.
* Their pain level will be more than 3 on visual analogue scale.
* Having mild to moderate score on Menstrual Distress questionnaire (MDQ) ( ≥ 50).
* Having regular menstruation for the last 6 months (every 28-30 days with no intermittent bleeding).

Exclusion Criteria:

* Systematic chronic diseases or any pelvic inflammatory diseases.
* Secondary dysmenorrhea.
* Menstrual irregularity.
* Nerve damage resulting in loss of feeling.
* Swelling, scar or skin infection.
* Diabetic patients.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessment | 3 months
  It will be assessed for each participant in both groups (A & B) before and after treatment, using the visual analogue scale (VAS). The VAS is usually presented as a 10 cm horizontal line on which the participants' pain intensity is represented by a point between the extremes of " no pain at all " and " worst pain imaginable ". It's simplicity, reliability and validity as well as its ratio scale properties make the VAS the optional tool for describing pain intensity.
Assessment of pain pressure threshold | 3 months
  A pressure algometer will be used to measure pain pressure thresholds (PPTs) for all participants in both groups before and after treatment, coinciding with peak menstrual pain on the first day of menstruation. Six specific points around the umbilicus and lower back will be assessed, with each point measured twice using a 1-cm² probe applied at 30kPa/s. The areas will be cleaned with alcohol before testing. Two points will be measured 4cm bilaterally from the umbilicus, two more 4cm below these, one 4cm below the umbilicus, and one in the lumbar region at S2-S4. The mean values of these points will be used for PPT data analysis.
Menstrual distress questionnaire (MDQ) | 3 months
  It will be used pre and post- treatment to assess the severity of symptoms of primary dysmenorrhea for all participants in both groups (A & B). The MDQ consists of symptoms or feelings associated with menstruation. The total number of items is 47. It is a 5 point rating scale from 0-4. For each items, there is 5 options i.e. No, mild, moderate, severe and very severe. An option of (very severe) has a score of 4, (severe) has a score of 3, (moderate) has a score of 2, (mild) has a score of 1, (No) has a score of 0. It includes seven sub-scales as (pain, water retention, autonomic reactions, negative affect, impaired concentration, mood and behavioral changes, arousal control). Overall Score was interpreted as follows :< 50 - mild , 50 to 70 - moderate and >70 severe.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Barmoud Nashed Kassab, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Doaa Ashraf Abd El-Ghany, Cairo, Egypt